CLINICAL TRIAL: NCT05067647
Title: A Prospective, Single-Arm Multi-Center Study of the ENSEAL® X1 Curved Jaw Tissue Sealer and Generator G11 in Thoracic, Urologic, and Ear, Nose, and Throat (ENT) Procedures
Brief Title: A Study of the ENSEAL® X1 Curved Jaw Tissue Sealer and Generator G11 in Thoracic, Urologic, and Ear, Nose, and Throat (ENT) Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG_2020_04; ENG_2020_04 (Other: Ethicon Endo-Surgery)
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Thoracic Procedure; Urologic Procedure; Ear, Nose and Throat Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Thoracic, Urologic, Ear, Nose and Throat (ENT) Procedures (Experimental): Any thoracic, urologic, or ENT procedure where ENSEAL X1 is used for transecting and sealing vessels according to instructions for use. Participants will be considered enrolled when the ENSEAL X1 device has been attempted to be used for a vessel transection during thoracic, urologic, or ENT procedures.
  Interventions: Device: ENSEAL X1 Curved Jaw Tissue Sealer

INTERVENTIONS:
Device: ENSEAL X1 Curved Jaw Tissue Sealer — ENSEAL X1 curved jaw tissue sealer is used for transecting and sealing vessels during thoracic, urologic, or ENT procedures according to instructions for use.

SUMMARY:
The purpose of this study is to demonstrate the acceptable performance and safety of the ENSEAL X1 curved jaw tissue sealer and Ethicon endo-surgery generator G11 (GEN11) devices when used per the instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

1. Primary laparoscopic or open procedure (thoracic, urologic or ear, nose, and throat [ENT]) where at least one vessel is planned to be transected by the ENSEAL X1 curved jaw tissue sealer (ENSEAL X1) device per the Instructions for use (IFU)
2. Willingness to give consent and comply with all study-related evaluations and treatment schedule
3. At least 18 years of age

Exclusion Criteria:

1. Physical or psychological condition which would impair study participation
2. Enrollment in a concurrent interventional clinical study that could impact the study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Endo-Surgery Clinical Trial, Study Director — Ethicon Endo-Surgery
Locations (6):
- Methodist Hospital, Omaha, Nebraska, United States
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - Kitasato University, Kanagawa
  - Kanagawa Cancer Center, Yokohama
- Zuyderland Medical Center, Sittard, Netherlands
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Siegel JM, Cummings JF, Clymer JW. Reproducible, repeatable and clinically-relevant hemostasis scoring. J Adv Med Pharm Sci 2014;1:30-39.

RESULTS

PARTICIPANT FLOW:
Groups:
- ENSEAL X1: All participants were treated with ENSEAL X1 device for transection of at least one vessel during thoracic, urologic, or ENT procedures.
Period: Overall Study
Arm/Group | ENSEAL X1
Started | 94
Completed | 93
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 61
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Vessels With Less Than or Equal to (<=) Grade 3 Hemostasis Based on Hemostasis Grading Scale
Description: A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with ENSEAL X1; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products). Here, the number of vessels that achieved <=Grade 3 hemostasis was reported.
Time Frame: On the day of transection (Day 0)
Population: ENSEAL X1 analysis set included all participants whose vessels were transected and analyzed during the procedures. Here, the number of vessels transected analyzed included all vessels that were transected and analyzed for this outcome measure.
Measure: Count of Units; unit: vessels transected
Units Other Than Participants: vessels transected
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 94
Number analyzed (vessels transected) | 112
vessels transected | 108

2. Primary Outcome: Number of Participants With at Least One Device-related Adverse Events (AEs)
Description: Device-related AEs were those having a relationship of possibly, probably, or causally. 1. Possible-The relationship with use of device was weak but cannot be ruled out completely. Alternative causes were also possible. Cases where relatedness cannot be assessed, or no information had been obtained were also classified as possible. 2. Probable -The relationship with use of device seemed relevant and/or event cannot reasonably be explained by another cause, but additional information may be obtained; 3. Causal relationship-The event was associated with device or with procedures beyond reasonable doubt with event occurred such as, a known side effect; temporal relationship; involves a body-site or organ that device was applied or had an effect on; followed a known response pattern; impact on event when discontinued and reintroduced; Others; Harms due to error in use.
Time Frame: Baseline up to 6 weeks
Population: ENSEAL X1 analysis set included all participants who utilized ENSEAL X1 device during the procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 94
Participants | 4

3. Secondary Outcome: Number of Participants With Adhesion Removal or Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for adhesion removal or division by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: ENSEAL X1 analysis set included all participants who utilized ENSEAL X1 device during the procedures. Here, the number of participants analyzed included participants who were analyzed only for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 13
Participants
  Very dissatisfied | 1
  Dissatisfied | 2
  Neither Satisfied or Dissatisfied | 0
  Satisfied | 6
  Very Satisfied | 4

4. Secondary Outcome: Number of Participants With Lymphatics Bundles Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for lymphatics bundles division by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 36
Participants
  Very dissatisfied | 1
  Dissatisfied | 1
  Neither Satisfied or Dissatisfied | 6
  Satisfied | 21
  Very Satisfied | 7

5. Secondary Outcome: Number of Participants With Tissue Bundles Division Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissue bundles division by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 57
Participants
  Very dissatisfied | 2
  Dissatisfied | 1
  Neither Satisfied or Dissatisfied | 10
  Satisfied | 33
  Very Satisfied | 11

6. Secondary Outcome: Number of Participants With Tissue Grasping Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissue grasping by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 27
Participants
  Very dissatisfied | 1
  Dissatisfied | 0
  Neither Satisfied or Dissatisfied | 3
  Satisfied | 13
  Very Satisfied | 10

7. Secondary Outcome: Number of Participants With Tissue Cutting Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissue cutting by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 58
Participants
  Very dissatisfied | 1
  Dissatisfied | 3
  Neither Satisfied or Dissatisfied | 6
  Satisfied | 39
  Very Satisfied | 9

8. Secondary Outcome: Number of Participants With Tissue Dissection Using ENSEAL X1 Device as Assessed by Surgeon Satisfaction Scale Score
Description: Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for tissue dissection by ENSEAL X1.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 52
Participants
  Very dissatisfied | 0
  Dissatisfied | 6
  Neither Satisfied or Dissatisfied | 8
  Satisfied | 31
  Very Satisfied | 7

9. Secondary Outcome: Number of Vessels With Hemostasis (Grade 1 to 4) Based on Grading Scale
Description: A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with ENSEAL X1; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products). Here, the number of vessels that achieved Grade 1 to 4 hemostasis was reported.
Time Frame: On the day of transection (Day 0)
Population: as for outcome 1
Measure: Count of Units; unit: vessels transected
Units Other Than Participants: vessels transected
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 94
Number analyzed (vessels transected) | 112
vessels transected
  Grade 1 | 104
  Grade 2 | 0
  Grade 3 | 4
  Grade 4 | 4

10. Secondary Outcome: Percentage of Grade 4 Vessel Transections Requiring Hemostasis Measures Such as Sutures and Hemoclips
Description: Percentage of grade 4 vessel transections requiring hemostasis measures such as sutures and hemoclips were reported.
Time Frame: On the day of transection (Day 0)
Population: ENSEAL X1 analysis set included all participants whose vessels were transected and analyzed during the procedures. Here, the number of participants analyzed included participants who were analyzed only for this outcome measure and the number of vessels transected analyzed included only vessels that were transected and analyzed for this outcome measure.
Measure: Number; unit: percentage of vessel transections
Units Other Than Participants: vessels transected
Arm/Group | ENSEAL X1
Number analyzed (Participants) | 4
Number analyzed (vessels transected) | 4
percentage of vessel transections
  Sutures | 50.0
  Hemoclips | 50.0

ADVERSE EVENTS:
Time Frame: Baseline up to 6 weeks
Description: ENSEAL X1 analysis set included all participants who utilized ENSEAL X1 device during the procedures.
Arm/Group | ENSEAL X1
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 4/94
Other Adverse Events (participants affected / at risk) | 22/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENSEAL X1 (N=94)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENSEAL X1 (N=94)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Ileus paralytic (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (6)
Catheter site extravasation (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 2 (2)
Suprapubic pain (General disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 1 (2)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7)
Wound complication (Injury, poisoning and procedural complications) | 9 (9)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 2 (2)
Blood albumin decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Oxygen consumption increased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2)
Urine output (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dizziness postural (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Venous haemorrhage (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT05067647/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT05067647/SAP_001.pdf